CLINICAL TRIAL: NCT06039670
Title: Percutaneous Transluminal Forceps Biopsy Combined With Transhepatic Biliary Drainage in the Management of Patients With Obstructive Jaundice: Efficacy, Safety and Accuracy
Brief Title: Percutaneous Transluminal Forceps Biopsy
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: PTFB
Record Dates: First submitted 2017-12-11; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-06

CONDITIONS: Biliary Stricture; Biopsy Wound; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: biliary biopsy — biliary biopsy through a percutaneous approach during a percutaneous biliary drainage

SUMMARY:
To evaluate during a 7 months period the efficacy, safety and accuracy of percutaneous transluminal forceps biopsy combined with transhepatic biliary drainage in patients with biliary stricture

DETAILED DESCRIPTION:
Biological parameters of liver function, histopathology of specimens, comparison with others clinical and pathological data (imaging follow up, percutaneous biopsy, surgical biopsy, endoscopic biopsy) were recorded Comparison between pathological findings of surgery or endoscopy or percutaneous biopsy and specimens coming from biliary forceps biopsy follow up of the patient 12 months after biopsy Evaluation of complications, accuracy

ELIGIBILITY:
Inclusion Criteria:

* Patients with biliary strictures without histology available

Exclusion Criteria:

* Pregnant patients
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with obstructive jaundice referred for percutaneous transhepatic biliary drainage without histological diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of PTBD | 7 days
  Efficacy of PTBD : bilirubinemia after PTFB at Day 7
accuracy for percutaneous biliary biopsy (PTFB) | from baseline up to 1 month
  Accuracy of PTFB : percentage of true positive and true negative results by pathologists
incidence of PTFB-related adverse events | up to 1 month after procedure
  Number of patients with PTFB related adverse-events as assessed by Society of Interventional Radiology Standards of Practice Committee classification

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Fohlen, Principal Investigator — Caen UH

IPD SHARING:
Plan to Share IPD: No